CLINICAL TRIAL: NCT00378092
Title: A Prospective Study of the Clinical Outcome Following Treatment Discontinuation After Remission in First-Episode Schizophrenia
Brief Title: A Follow-Up Study of Schizophrenic Participants Following Treatment Discontinuation After Remission From a First Psychotic Episode
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Cilag N.V./S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR011992; RISSCH3024
Record Dates: First submitted 2006-09-15; First posted 2006-09-19 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-05

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Risperidone; Risperdal consta
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Risperidone Long-Acting Injection (RLAI) (Period 1) (Experimental): Participants will receive 25 milligram (mg) to 50 mg of RLAI intramuscularly (into the muscle) which will be tapered and discontinued over a period of up to 6 weeks. Participants will be followed-up until their first disease relapse or maximum of 36 months.
  Interventions: Drug: Risperidone Long-Acting Injection (RLAI)
- Oral risperidone and RLAI (Period 2) (Experimental): Participants who will experience a disease relapse, will receive RLAI 25 mg, 37.5 mg, or 50 mg, every 2 weeks as an intramuscular injection in the gluteus (a muscle) for up to 24 months. Supplementation with oral risperidone 1 mg or 2 mg or 3 mg will be administered for 21 days from the first dose of RLAI (until RLAI injections becomes effective) and then taper off over the next 5 days. Thereafter, oral risperidone can be administered at the discretion of the Investigator if additional antipsychotic medication will be required due to acute exacerbation of symptoms between visits.
  Interventions: Drug: Oral risperidone; Drug: Risperidone Long-Acting Injection (RLAI)

INTERVENTIONS:
Drug: Oral risperidone — Oral risperidone 1 mg or 2 mg or 3 mg will be administered for 21 days from the first dose of RLAI (until RLAI injection becomes effective) and then taper off over the next 5 days. Thereafter, oral risperidone can be administered at the discretion of the Investigator if additional antipsychotic medication will be required due to acute exacerbation of symptoms between visits.
  Arms: Oral risperidone and RLAI (Period 2)
Drug: Risperidone Long-Acting Injection (RLAI) — RLAI 25 mg to 50 mg will be administered, intramuscularly which will be tapered and discontinued over a period of up to 6 weeks.
  Other Names: Risperdal consta
  Arms: Risperidone Long-Acting Injection (RLAI) (Period 1)
Drug: Risperidone Long-Acting Injection (RLAI) — Participants who will experience a disease relapse, will receive RLAI 25 mg, 37.5 mg, or 50 mg, every 2 weeks as an intramuscular injection in the gluteus for up to 24 months.
  Other Names: Risperdal consta
  Arms: Oral risperidone and RLAI (Period 2)

SUMMARY:
The purpose of this study is to evaluate the outcome of medication discontinuation, the safety and effectiveness of re-initiating risperidone long acting injection (RLAI) in case of relapse (the return of a medical problem) of schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality, often with delusions and hallucinations, and withdrawal into the self) during the study observation period of 36 months.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), prospective (study following participants forward in time), single-arm, single-center study to assess the consequences of treatment discontinuation and evaluate clinical response to re-initiation of risperidone in case of relapse. The study will consist of 2 periods: Period 1 and Period 2. Participants who were on RLAI for 24 months and in remission (when a medical problem gets better or goes away at least for a while) state will enter in Period 1. In Period 1: RLAI will be tapered and discontinued over a period of 6 weeks. Participants will be regularly and carefully followed-up until their first disease relapse or a maximum of 36 months. In case of relapse (i.e., participants experience the same or similar symptoms to those experienced at the time of study entry in the previous Study RIS-PSY-301), participants will be transferred from Period 1 to Period 2. In Period 2, participants will re-start medication with RLAI (25 milligram [mg], 37.5 mg, or 50 mg [maximum]) and simultaneously start on oral (taken by mouth) risperidone (1 mg, 2 mg, or 3 mg). Doses will be adjusted at Investigator's discretion. Oral Risperidone will only be given for the first 3 weeks until the RLAI injection becomes effective. RLAI injections will continue for up to a maximum of 24 months. Participants will be followed-up until a (new) relapse or the treatment stopped, during a maximum of 24 months. The total duration of the study will be 36 months and will include 16 visits. Assessments will be performed every 2 months in the first year and every 3 months during the following 24 months period. Time to relapse and rate of relapse will be measured as primary outcome for Period 1 and degree of clinical improvement will be measured by Positive And Negative Syndrome Scale (PANSS) total score for schizophrenia. Time to response after re-exposure to treatment with RLAI will be measured as primary outcome for Period 2. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria: - Participants who completed 24 months RIS-PSY-301 study - Surgically sterile female participants or practicing an effective method of birth control before entry and throughout the study; and must have shown a negative urine serum pregnancy test at baseline before study entry - Participants who have signed informed consent document Exclusion Criteria: - Participants requiring treatment with mood stabilizers or antidepressants at study entry - Participants with evidence of alcohol or drug abuse or dependence (except for nicotine and caffeine dependence) according to Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria diagnosed in the last month before entry - Participants with a history of severe drug allergy, drug hypersensitivity, or neuroleptic malignant (cancerous) syndrome - Participants with known hypersensitivity to risperidone - Participants with acute risk of suicide at study entry or a history of suicidal attempt(s)

Ages: 17 Years to 47 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2006-04; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Time to Relapse After Discontinuation of Risperidone Long-Acting Injection (RLAI) in First-Episode Participants Successfully Treated for 24 Months With RLAI in Previous Study (RIS-PSY-301) (Period 1) | Month 36 or early withdrawal (EW)
  Relapse will be diagnosed if 1 or more of the following occurs: a 25 percent increase in Positive and Negative Syndrome Scale (PANSS) total score ranging from 30 (absent) to 210 (extreme ill); Clinical Global Impression (CGI-C) score of 6 ('much worse'); deliberate self-injury (as per adverse event [AE] reporting); emergence of clinically significant suicidal or homicidal ideation (as per AE reporting); or violent behavior resulting in significant injury to another person or significant property damage (as per AE reporting).
Percentage of Participants who Relapsed After Discontinuation of RLAI (Period 1) | Month 36 or EW
  Relapse will be diagnosed if 1 or more of the following occurs: a 25 percent increase in PANSS total score ranging from 30 (absent) to 210 (extreme ill); CGI-C score of 6 ('much worse'); deliberate self-injury (as per AE reporting); emergence of clinically significant suicidal or homicidal ideation (as per AE reporting); or violent behavior resulting in significant injury to another person or significant property damage (as per AE reporting).
Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score After Re-Initiation of RLAI, at Month 24 or EW (Period 2) | Baseline and Month 24 or EW
  The PANSS is a medical scale that assesses various symptoms of schizophrenia and provides a total score (sum of the scores of all 30 items) and scores for 3 subscales: positive subscale (7 items), negative subscale (7 items), and general psychopathology subscale (16 items), each rated on a scale of 1 (absent) to 7 (extreme). The total score is the sum of all 30 PANSS items, with a range of 30 (absent) to 210 (extreme ill). Higher scores indicate worsening.
Time to Treatment Response After Re-Initiation of RLAI (Period 2) | Month 24 or EW
  Time to treatment response after re-initiation of RLAI will be the time that elapse between Baseline assessment of PANSS for Period 2 and fulfilment of the response which is defined as greater than or equal to 20 percent improvement in PANSS total score. PANSS is a medical scale that assesses various symptoms of schizophrenia and provides a total score (sum of the scores of all 30 items) with a range of 30 (absent) to 210 (extreme ill). Higher scores indicate worsening.

SECONDARY OUTCOMES:
Change From Baseline in PANSS Total Score and Subscales of PANSS at Month 36 or EW (Period 1) | Baseline and Month 36 or EW
  The PANSS is a medical scale that assesses various symptoms of schizophrenia and provides a total score (sum of the scores of all 30 items) and scores for 3 subscales: positive subscale (7 items), negative subscale (7 items), and general psychopathology (GP) subscale (16 items), each rated on a scale of 1 (absent) to 7 (extreme). The total score is the sum of all 30 PANSS items, with a range of 30 (absent) to 210 (extreme ill). Higher scores indicate worsening.
Change From Baseline in PANSS Total Score and Subscales of PANSS at Month 24 or EW (Period 2) | Baseline and Month 24 or EW
  The PANSS is a medical scale that assesses various symptoms of schizophrenia and provides a total score (sum of the scores of all 30 items) and scores for 3 subscales: positive subscale (7 items), negative subscale (7 items), and general psychopathology (GP) subscale (16 items), each rated on a scale of 1 (absent) to 7 (extreme). The total score is the sum of all 30 PANSS items, with a range of 30 (absent) to 210 (extreme ill). Higher scores indicate worsening.
Change From Baseline in Marder PANSS Subscales Score at Month 36 or EW (Period 1) | Baseline and Month 36 or EW
  The PANSS total score consists of the sum of all 30 PANSS items and score ranges from 30 to 210. Higher scores indicate worsening. The symptoms are rated on a 7-point Marder scale from 1 (absent) to 7 (extreme psychopathology). Positive symptoms subscale consists of 8 items with total score range of 856; negative symptoms subscale and disorganized thoughts subscale, each consists of 7 items with total score range of 7-49, uncontrolled hostility (UH) or excitement subscale and anxiety/depression subscale, each consists of 4 items with total score range of 4-28.
Change From Baseline in Marder PANSS Subscales Score at Month 24 or EW (Period 2) | Baseline and Month 24 or EW
  The PANSS is a 30-item scale to assess the neuropsychiatric symptoms of schizophrenia. The symptoms are rated on a 7-point Marder scale from 1 (absent) to 7 (extreme psychopathology). Positive symptoms subscale consists of 8 items with total score range of 8-56; negative symptoms subscale and disorganized thoughts subscale, each consists of 7 items with total score range of 7-49, UH or excitement subscale and anxiety or depression subscale, each consists of 4 items with total score range of 4-28. Higher score indicates greater severity.
Number of Participants With Disease Remission Based on PANSS (Period 1) | Month 36 or EW
  A participants will be 'in remission' when he/she is symptomatically stable and show progressive improvement in total recovery according to severity (mild or less simultaneously on 8 PANSS items:P1 delusions, P2 conceptual disorganization, P3 hallucinatory behavior, G9 unusual thought content, G5 mannerisms and posturing, N1 blunted affect, N4 social withdrawal, N6 lack of spontaneity or flow of conversation) and time (scores for 8 PANSS items above should not exceed the severity criterion mild at any time point of assessment for at least 6 months to meet the criteria of remission) criteria.
Number of Participants With Disease Remission Based on PANSS (Period 2) | Month 24 or EW
  A participants will be 'in remission' when he/she is symptomatically stable and show progressive improvement in total recovery according to severity (mild or less simultaneously on 8 PANSS items:P1 delusions, P2 conceptual disorganization, P3 hallucinatory behavior, G9 unusual thought content, G5 mannerisms and posturing, N1 blunted affect, N4 social withdrawal, N6 lack of spontaneity or flow of conversation) and time (scores for 8 PANSS items above should not exceed the severity criterion mild at any time point of assessment for at least 6 months to meet the criteria of remission) criteria.
Change From Baseline in Clinical Global Impression of Severity (CGI-S) Score at Month 36 or EW (Period 1) | Baseline and Month 36 or EW
  The CGI-S scale is a 7-point global assessment that measures the Clinician's impression of the severity of illness exhibited by a participant. A rating of '1=Normal, not at all ill' and a rating of '7=Among the most extremely ill participants'. Higher scores indicate worsening.
Clinical Global Impression of Change (CGI-C) Score at Month 36 or EW (Period 1) | Month 36 or EW
  The CGI-C scale is designed to assess the change in the clinical condition over time. The CGI-C consists of a 7-point rating of change, questioning if the clinical condition of the participant improved, remained unchanged, or worsened.
Change From Baseline in Clinical Global Impression of Severity (CGI-S) Score at Month 24 or EW (Period 2) | Baseline and Month 24 or EW
  The CGI-S scale is a 7-point global assessment that measures the Clinician's impression of the severity of illness exhibited by a participant. A rating of '1=Normal, not at all ill' and a rating of '7=Among the most extremely ill participants'. Higher scores indicate worsening.
Clinical Global Impression of Change (CGI-C) Score in Period 2 at Month 24 or EW (Period 2) | Month 24 or EW
  The CGI-C scale is designed to assess the change in the clinical condition over time. The CGI-C consists of a 7-point rating of change, questioning if the clinical condition of the participant improved, remained unchanged, or worsened.
Change From Baseline in Calgary Depression Scale Score for Schizophrenia (CDSS) at Month 36 or EW (Period 1) | Baseline and Month 36 or EW
  The CDSS assesses the level of depression in participants with schizophrenia. It consists of 9 items: depression, hopelessness, self-depreciation, pathological guilt, guilty ideas of reference, morning depression, early awakening, suicidal, observed depression, each scored on a 4-point scale (0=absent, 1=mild, 2=moderate, 3=severe). The total score is a sum of the scores of each item and may range from 0 to 27. Higher score indicates more severe pathology.
Change From Baseline in Calgary Depression Scale Score for Schizophrenia (CDSS) at Month 24 or EW (Period 2) | Baseline and Month 24 or EW
  The CDSS assesses the level of depression in participants with schizophrenia. It consists of 9 items: depression, hopelessness, self-depreciation, pathological guilt, guilty ideas of reference, morning depression, early awakening, suicidal, observed depression, each scored on a 4-point scale (0=absent, 1=mild, 2=moderate, 3=severe). The total score is a sum of the scores of each item and may range from 0 to 27. Higher score indicates more severe pathology.
Change From Baseline in Social and Occupational Functioning Assessment Scale (SOFAS) Score at Month 36 or EW (Period 1) | Baseline and Month 36 or EW
  The SOFAS is a 100- point single item scale that assesses level of social and occupational functioning of a participant and is not directly influenced by the overall severity of the individual's psychological symptoms.The scale values range from 1=most impaired to 100=healthiest individual. The scale also includes a rating point of 0=missing information.
Change From Baseline in Social and Occupational Functioning Assessment Scale (SOFAS) Score at Month 24 or EW (Period 2) | Baseline and Month 24 or EW
  The SOFAS is a 100-point single item scale that assesses level of social and occupational functioning of a participant and is not directly influenced by the overall severity of the individual's psychological symptoms.The scale values range from 1=most impaired to 100=healthiest individual. The scale also includes a rating point of 0=missing information.
Change From Baseline in Patient Global Impression-Severity (PGI-S) Score at Month 36 or EW (Period 1) | Baseline and Month 36 or EW
  The PGI-S is an 11-point (0=very well to 10=very poor) scale that requires the participants to rate the severity of their illness at the time of assessment, relative to the participant's past experience. The response options are: very much improved; much improved; improved (just enough to make a difference); no change; worse (just enough to make a difference); much worse; or very much worse.
Patient Global Impression-Change (PGI-C) Score at Month 36 or EW (Period 1) | Month 36 or EW
  The PGI-C is a 7-point scale that requires the participants to assess how much their illness has improved or worsened relative to a baseline state at the beginning of the intervention. The response options are: very much improved; much improved; improved (just enough to make a difference); no change; worse (just enough to make a difference); much worse; or very much worse .
Change From Baseline in Patient Global Impression-Severity (PGI-S) Score at Month 24 or EW (Period 2) | Baseline and Month 24 or EW
  The PGI-S is an 11-point (0=very well to 10=very poor) scale that requires the participants to rate the severity of their illness at the time of assessment, relative to the participant's past experience. The response options are: very much improved; much improved; improved (just enough to make a difference); no change; worse (just enough to make a difference); much worse; or very much worse.
Patient Global Impression-Change (PGI-C) Score at Month 24 or EW (Period 2) | Month 24 or EW
  The PGI-C is a 7-point scale that requires the participants to assess how much their illness has improved or worsened relative to a baseline state at the beginning of the intervention. The response options are: very much improved; much improved; improved (just enough to make a difference); no change; worse (just enough to make a difference); much worse; or very much worse .
Change From Baseline in 12-Item Short-Form (SF-12) Score - Quality of Life Survey at Month 36 or EW (Period 1) | Baseline and Month 36 or EW
  The SF-12 is a validated 12 question quality-of-life questionnaire. The SF-12 extracts 12 items from the SF-36 questionnaire in 2 six-item subscales: physical component summary (PCS) and MCS (mental component summary). The SF-12 score ranges from 10=maximum impairment to 70=no impairment.
Change From Baseline in 12-Item Short-Form (SF-12) Score - Quality of Life Survey at Month 24 or EW (Period 2) | Baseline and Month 24 or EW
  The SF-12 is a validated 12 question quality-of-life questionnaire. The SF-12 extracts 12 items from the SF-36 questionnaire in 2 six-item subscales: physical component summary (PCS) and MCS (mental component summary). The SF-12 scores range from 10=maximum impairment to 70=no impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag N.V./S.A., Belgium Clinical Trial, Study Director — Janssen Cilag N.V./S.A.
Locations (1):
- Bellville, South Africa

REFERENCES:
- [Derived] Emsley R, Oosthuizen PP, Koen L, Niehaus DJ, Martinez G. Symptom recurrence following intermittent treatment in first-episode schizophrenia successfully treated for 2 years: a 3-year open-label clinical study. J Clin Psychiatry. 2012 Apr;73(4):e541-7. doi: 10.4088/JCP.11m07138. PMID 22579160
- See also: Follow up of Schizophrenic Patients Following Treatment Discontinuation After Remission From a First Psychotic Episode — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=248&filename=CR011992_CSR_synopsis.pdf